CLINICAL TRIAL: NCT06521138
Title: The Effect of Transtheoretical Model-Based Antenatal and Postnatal Motivational Interviewing on Contraceptive Self-Efficacy, Contraceptive Attitude and Contraceptive Use: A Randomized Controlled Trial
Brief Title: The Effect of Transtheoretical Model-Based Motivational Interviewing on Postpartum Contraception
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Aliye DOĞAN GANGAL, Principal Investigator, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 711519
Record Dates: First submitted 2024-07-16; First posted 2024-07-25 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Supportive Care
Keywords: contraception; family planning; contraceptive self efficacy; contraceptive attitude; postpartum contraception
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinding of the outcome assessors in this study was planned. The data obtained from the research will be coded as A and B by an independent researcher and transferred to the SPSS program. The data will be analyzed by an independent statistical expert.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational interviewing group (Experimental): Antenatal and postnatal motivational interviewing based on the transtheoretical model will be applied.
  Interventions: Behavioral: Motivational interviewing group
- Control group (Other): The control group receiving routine care.
  Interventions: Other: Control group

INTERVENTIONS:
Behavioral: Motivational interviewing group — The intervention group will receive motivational interviewing based on the transtheoretical model in addition to routine care. Motivational interviews are structured in line with the stages of change and behavioral change processes, which are the basic structures of the transtheoretical model. Three sessions of motivational interviewing with a session duration of 30 min will be implemented. Two sessions of motivational interviewing in the prenatal period and one session of motivational interviewing in the postnatal period.
  Other Names: Transtheoretical model-based motivational interviewing group
  Arms: Motivational interviewing group
Other: Control group — Participants in the control group will receive routine care at the center.
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to evaluate the effect of transtheoretical model-based antenatal and postnatal motivational interviewing on contraceptive self-efficacy, contraceptive attitude, and postpartum contraception use. This study was planned as a single-centre, parallel-group, randomized controlled trial design. The study group consisted of 72 women at 28-32 weeks of gestation (intervention group n=36, control group n=36). Block randomization stratified by parity will be used to assign participants to groups. The intervention group will receive antenatal and postnatal motivational interviewing in addition to routine care, while the control group will receive routine care only. Outcomes will be evaluated at 12 weeks postpartum. Data will be collected using a personal information form, Contraceptive Self-Efficacy Scale, Contraceptive Attitude Questionnaire, Contraceptive Use Form and Stages of Behavior Change Short Form.

DETAILED DESCRIPTION:
Short gestational intervals are known to be directly associated with adverse pregnancy outcomes, such as gestational diabetes, maternal obesity, anemia, maternal mortality, severe maternal morbidity, preterm delivery, low birth weight, and infant mortality. The most important step in establishing optimum pregnancy intervals can be achieved by meeting the contraceptive needs of postpartum women. Motivational interviewing incorporates components of contraception counseling best practices, such as building trust, optimizing the decision-making process, improving self-efficacy, and protecting the autonomy of the individual, which allows it to be actively used in the counseling process. Therefore, this study aimed to investigate the effects of transtheoretical model-based motivational interviewing on postpartum contraception. In this study, the intervention group will receive two motivational counseling sessions in the antenatal period and one motivational interviewing session in the postnatal period in addition to routine care, while the control group will receive only routine care. The data will be coded as A and B in SPSS (Statistical Package for the Social Sciences) and analyzed by an independent statistical expert.

ELIGIBILITY:
Inclusion Criteria:

* 28 to 32 weeks of gestation
* At least literate in Turkish
* Agree to participate in the study
* Willing to participate in the postpartum follow-up
* Having access to a smartphone

Exclusion Criteria:

* Women who do not have a sexual partner
* Women who give consent for female sterilization immediately after delivery

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — The sample of this study consists of pregnant women.
Enrollment: 72 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Postpartum contraceptive method use questionnaire | 12 weeks postpartum
  The questionnaire assesses the contraceptive method used by the participants in the postpartum period. It consist of questions assessing the contraceptive method used by the participants and the time of onset. The number of participants using modern contraceptive methods in the postpartum period has been reported.
Contraceptive Attitude Questionnaire | At baseline and 12 weeks postpartum
  It was developed to assess contraceptive attitude. Contraceptive attitude questionnaire consists of three sub-dimensions ; effects on family economy and sexual life, effects on moral values of the society, effects on men and religion. The higher the score, the higher the contraceptive attitude.
Contraceptive Self Efficacy Scale | At baseline and 12 weeks postpartum
  Women's contraceptive self-efficacy will be assessed using the Turkish version of the Contraceptive Self-Efficacy Scale. The scale consists of 11 items and three sub-dimensions; (1) husband/partner communication, (2) provider communication, (3) choosing and managing a method. The total score ranged from 0 to 110. Higher scores indicate higher levels of contraceptive self-efficacy.

SECONDARY OUTCOMES:
Stages of Behavior Change | At baseline and 12 weeks postpartum
  The transtheoretical model (stages of change model), which is widely used to determine the process of behavior change, was adapted to postpartum contraception behavior. This form will be used to assess participants' stages of behavior change (precontemplation, contemplation, preparation, action, maintenance) regarding contraceptive use.

CONTACTS AND LOCATIONS:
Overall Officials: Aliye Dogan Gangal, Principal Investigator — Gazi University
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There are no plans to make individual participant data available to other researchers.

REFERENCES:
- [Background] Bergo CJ, Handler A, Geller S, Grobman WA, Awadalla S, Rankin K. Interpregnancy Interval and Severe Maternal Morbidity in Iowa, 2009 to 2014. Womens Health Issues. 2021 Sep-Oct;31(5):503-509. doi: 10.1016/j.whi.2021.04.005. Epub 2021 Jun 1. PMID 34088600
- [Background] Ball SJ, Pereira G, Jacoby P, de Klerk N, Stanley FJ. Re-evaluation of link between interpregnancy interval and adverse birth outcomes: retrospective cohort study matching two intervals per mother. BMJ. 2014 Jul 23;349:g4333. doi: 10.1136/bmj.g4333. PMID 25056260
- [Background] Hutcheon JA, Nelson HD, Stidd R, Moskosky S, Ahrens KA. Short interpregnancy intervals and adverse maternal outcomes in high-resource settings: An updated systematic review. Paediatr Perinat Epidemiol. 2019 Jan;33(1):O48-O59. doi: 10.1111/ppe.12518. Epub 2018 Oct 12. PMID 30311955
- [Background] ACOG Committee Opinion No. 736: Optimizing Postpartum Care. Obstet Gynecol. 2018 May;131(5):e140-e150. doi: 10.1097/AOG.0000000000002633. PMID 29683911
- [Background] American College of Obstetricians and Gynecologists; Society for Maternal-Fetal Medicine. Obstetric Care Consensus No. 8: Interpregnancy Care. Obstet Gynecol. 2019 Jan;133(1):e51-e72. doi: 10.1097/AOG.0000000000003025. PMID 30575677
- [Background] Dev R, Kohler P, Feder M, Unger JA, Woods NF, Drake AL. A systematic review and meta-analysis of postpartum contraceptive use among women in low- and middle-income countries. Reprod Health. 2019 Oct 29;16(1):154. doi: 10.1186/s12978-019-0824-4. PMID 31665032
- [Background] Brunson MR, Klein DA, Olsen CH, Weir LF, Roberts TA. Postpartum contraception: initiation and effectiveness in a large universal healthcare system. Am J Obstet Gynecol. 2017 Jul;217(1):55.e1-55.e9. doi: 10.1016/j.ajog.2017.02.036. Epub 2017 Feb 28. PMID 28257962
- [Background] Wakuma B, Mosisa G, Etafa W, Mulisa D, Tolossa T, Fetensa G, Besho M, Gebre M, Tsegaye R. Postpartum modern contraception utilization and its determinants in Ethiopia: A systematic review and meta-analysis. PLoS One. 2020 Dec 14;15(12):e0243776. doi: 10.1371/journal.pone.0243776. eCollection 2020. PMID 33315904
- [Background] Lopez LM, Grey TW, Tolley EE, Chen M. Brief educational strategies for improving contraception use in young people. Cochrane Database Syst Rev. 2016 Mar 30;3(3):CD012025. doi: 10.1002/14651858.CD012025.pub2. PMID 27027480
- [Background] Zapata LB, Murtaza S, Whiteman MK, Jamieson DJ, Robbins CL, Marchbanks PA, D'Angelo DV, Curtis KM. Contraceptive counseling and postpartum contraceptive use. Am J Obstet Gynecol. 2015 Feb;212(2):171.e1-8. doi: 10.1016/j.ajog.2014.07.059. Epub 2014 Aug 2. PMID 25093946
- [Background] Cavallaro FL, Benova L, Owolabi OO, Ali M. A systematic review of the effectiveness of counselling strategies for modern contraceptive methods: what works and what doesn't? BMJ Sex Reprod Health. 2020 Oct;46(4):254-269. doi: 10.1136/bmjsrh-2019-200377. Epub 2019 Dec 11. PMID 31826883
- [Background] Engelbert Bain L, Amu H, Enowbeyang Tarkang E. Barriers and motivators of contraceptive use among young people in Sub-Saharan Africa: A systematic review of qualitative studies. PLoS One. 2021 Jun 4;16(6):e0252745. doi: 10.1371/journal.pone.0252745. eCollection 2021. PMID 34086806
- [Background] Wilson A, Nirantharakumar K, Truchanowicz EG, Surenthirakumaran R, MacArthur C, Coomarasamy A. Motivational interviews to improve contraceptive use in populations at high risk of unintended pregnancy: a systematic review and meta-analysis. Eur J Obstet Gynecol Reprod Biol. 2015 Aug;191:72-9. doi: 10.1016/j.ejogrb.2015.05.010. Epub 2015 Jun 11. PMID 26093351
- [Background] Rodriguez J, Abutouk M, Roque K, Sridhar A. Personalized contraceptive counseling: helping women make the right choice. Open Access J Contracept. 2016 May 11;7:89-96. doi: 10.2147/OAJC.S81546. eCollection 2016. PMID 29386940
- [Background] Gregory EF, Maddox AI, Levine LD, Fiks AG, Lorch SA, Resnicow K. Motivational interviewing to promote interconception health: A scoping review of evidence from clinical trials. Patient Educ Couns. 2022 Nov;105(11):3204-3212. doi: 10.1016/j.pec.2022.07.009. Epub 2022 Jul 16. PMID 35870992
- [Background] Frost H, Campbell P, Maxwell M, O'Carroll RE, Dombrowski SU, Williams B, Cheyne H, Coles E, Pollock A. Effectiveness of Motivational Interviewing on adult behaviour change in health and social care settings: A systematic review of reviews. PLoS One. 2018 Oct 18;13(10):e0204890. doi: 10.1371/journal.pone.0204890. eCollection 2018. PMID 30335780
- [Background] Whiting-Collins L, Grenier L, Winch PJ, Tsui A, Donohue PK. Measuring contraceptive self-efficacy in sub-Saharan Africa: development and validation of the CSESSA scale in Kenya and Nigeria. Contracept X. 2020 Oct 9;2:100041. doi: 10.1016/j.conx.2020.100041. eCollection 2020. PMID 33145490